CLINICAL TRIAL: NCT01890421
Title: Multicenter Open-label Study to Evaluate Efficacy of Gadobutrol-enhanced Cardiac Magnetic Resonance Imaging (CMRI) for Detection of Significant Coronary Artery Disease (CAD) in Subjects With Known or Suspected CAD by a Blinded Image Analysis
Brief Title: Gadobutrol/Gadavist-enhanced Cardiac Magnetic Resonance Imaging (CMRI) to Detect Coronary Artery Disease (CAD)
Acronym: GadaCAD 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15961; 2012-002563-10 (EudraCT Number)
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Perfusion Imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gadobutrol 0.1 mmol/kg body weight (Experimental): Participants received gadobutrol at the total approved standard dose of 0.1 millimole per kilogram body weight (mmol/kg BW) in 2 separate bolus injections: 0.05 mmol/kg BW at peak pharmacologic stress and 0.05 mmol/kg BW at rest via a power injector.
  Interventions: Drug: Gadobutrol (Gadovist, Gadavist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, Gadavist, BAY86-4875) — Participants received gadobutrol at the total approved standard dose of 0.1 millimole per kilogram body weight (mmol/kg BW) in 2 separate bolus injections: 0.05 mmol/kg BW at peak pharmacologic stress and 0.05 mmol/kg BW at rest via a power injector.

SUMMARY:
Participants being evaluated for suspected or known Coronary artery Disease (CAD) based on signs and/or symptoms, will be invited to participate in the study. The duration for a participant in the study may range from 2 days to 4-6 weeks. One to four visits to the study doctor will be required.

This study will investigate the diagnostic results of gadobutrol-enhanced Cardiac Magnetic Resonance Imaging (CMRI) images regarding the detection (sensitivity) and exclusion (specificity) of coronary artery disease utilizing a uniform image acquisition software. The CMR images will be tested either against the results from routine clinical Coronary Angiography (CA) or those from Computed Tomography Angiography (CTA), which is used as the standard of reference. The CA/CTA may have been performed up to 4 weeks prior to enrollment or be scheduled up to 4/6 weeks after the study.

CMRI and CA/CTA images will be collected for an independent image review (blinded read).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years
* Participants with suspected or known CAD based on signs and/or (typical or atypical) chest pain who have routine CA without intervention or CTA within 4 weeks around gadobutrol-enhanced CMRI
* Willingness to undergo stress/rest CMRI and to follow directions and complete all study procedures
* Women of childbearing potential (e.g. age < 60y, no history of surgical sterilization or hysterectomy): use of contraception and a negative pregnancy test

Exclusion Criteria:

* Suspected clinical instability or unpredictability of the clinical course during the study period
* Contraindication to the cardiac MRI examination (e.g. inability to hold breath; severe claustrophobia, metallic devices such as pace makers)
* History of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents according to the investigator's assessment / judgment
* Estimated glomerular filtration rate (eGFR) value <30 mL/min/1.73 m^2 derived from a serum / blood creatinine result within 2 weeks prior to gadobutrol injection. Any participant on hemodialysis or peritoneal dialysis is excluded from enrollment.
* Acute renal insufficiency
* Coronary artery bypass grafting (CABG)
* Acute myocardial infarction (< 14 days prior to inclusion), unstable angina / acute coronary syndrome, severe congestive heart failure
* Irregular heart rhythm
* Condition that precludes the safe administration of pharmacological stressor according to the respective approved label such as sinus node disease, 2nd or 3rd degree atrioventricular block, obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2013-07-19 (Actual); Primary Completion 2015-04-10 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Minneapolis, Minnesota, United States
- France (2):
  - Marseille
  - Saint-Etienne
- Germany (9):
  - Bad Krozingen, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Darmstadt, Hesse
  - Göttingen, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Leipzig, Saxony
  - Berlin
- Auckland, New Zealand
- South Korea (3):
  - Incheon
  - Seoul
  - Yangsan
- Lugano, Canton Ticino, Switzerland
- United Kingdom (3):
  - Leicester
  - Liverpool
  - London

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 study centers in 7 countries (Germany, South Korea, United Kingdom, France, United States, New Zealand and Switzerland), between 19 July 2013 (first subject first visit) and 10 April 2015 (last subject last visit).
Pre-assignment Details: Overall, 456 participants signed the informed consent, of them 19 did not finish their baseline visit (6 screening failure, 13 dropped out), 1 discontinued the study due to an adverse event (AE). A total of 436 participants entered the diagnostic imaging phase, of them 426 were treated with gadobutrol and entered the follow-up phase.
Period: Overall Study
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Started | 426
Completed | 415
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Other reason | 10

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF)
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 426
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 414
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 111
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 310
  More than one race | 0
  Unknown or Not Reported | 3
Childbearing Potential [Number; unit: Count of Participants]
  Of childbearing potential (only females) | 20
  No childbearing potential (only females) | 109
  No childbearing potential (only males) | 297
Body Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 79.75 (16.29)
Height [Mean (Standard Deviation); unit: Centimeter] | 170.99 (9.17)
Body Mass Index [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 27.160 (4.561)
Country [Count of Participants; unit: Participants]
  Germany | 210
  South Korea | 108
  Switzerland | 44
  United States of America | 31
  United Kingdom | 28
  France | 4
  New Zealand | 1
Age Categorical [Number; unit: Count of Participants]
  < 45 years | 60
  >= 45 to <= 64 years | 232
  >= 65 years | 134
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR (based on serum/blood creatinine from local laboratory) was measured/evaluated within 2 weeks before the first gadobutrol injection (at the latest on the day of gadobutrol-enhanced CMRI before the first gadobutrol injection).
  mL/min/1.73m^2 | 84.2 (18.37)

OUTCOME MEASURES:

1. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI (Based on RPS) - Primary Analysis of Sensitivity Based on Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=50% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 minute (min) post-injection
Population: Full analysis set (FAS): participants who underwent pharmacologic stress and for whom electronic case report form entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for SoR diagnosis were available. N=FAS with significant CAD (defined as maximum stenosis severity of >=50% by QCA) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 141
Sensitivity %
  Reader 1 | 76.6 [68.7 to 83.3]
  Reader 2 | 65.2 [56.8 to 73.1]
  Reader 3 | 64.5 [56.0 to 72.4]

2. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI (Based on RPS) - Additional Secondary Analysis of Sensitivity Based on the Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=70% for secondary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: FAS: participants who underwent pharmacologic stress and for whom electronic case report form (eCRF) entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for SoR diagnosis were available. N=FAS with significant CAD (defined as maximum stenosis severity of >=70% by QCA) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 108
Sensitivity %
  Reader 1 | 89.8 [82.5 to 94.8]
  Reader 2 | 79.6 [70.8 to 86.8]
  Reader 3 | 78.7 [69.8 to 86.0]

3. Primary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI (Based on RPS) - Primary Analysis of Specificity Based on the Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=50% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR). Specificity= true negative/ (true negative + false positive).
Time Frame: 0 to 30/40 min post-injection
Population: FAS included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for SoR diagnosis were available. N=FAS participants with significant CAD (defined as maximum stenosis severity of >=50% by QCA) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 235
Specificity %
  Reader 1 | 85.1 [79.9 to 89.4]
  Reader 2 | 92.3 [88.2 to 95.4]
  Reader 3 | 91.9 [87.7 to 95.1]

4. Primary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI (Based on RPS) - Additional Secondary Analysis of Specificity Based on the Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=70% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR). Specificity= true negative/ (true negative + false positive). This additional secondary analysis of specificity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: FAS included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for SoR diagnosis were available. N=FAS participants with significant CAD (defined as maximum stenosis severity of >=70% by QCA) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 268
Specificity %
  Reader 1 | 82.8 [77.8 to 87.2]
  Reader 2 | 91.0 [87.0 to 94.2]
  Reader 3 | 90.7 [86.5 to 93.9]

5. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Primary Analysis of Sensitivity Comparison Based on the Blinded Readers' Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by blinded readers' assessment. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=50% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 141
Sensitivity %
  Gadobutrol-enhanced CMRI-Reader 1 | 76.6
  Gadobutrol-enhanced CMRI-Reader 2 | 65.2
  Gadobutrol-enhanced CMRI-Reader 3 | 64.5
  Unenhanced CMRI-Reader 1 | 77.3
  Unenhanced CMRI-Reader 2 | 36.2
  Unenhanced CMRI-Reader 3 | 40.4
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 1 for presence of a myocardial perfusion defect indicating significant cad per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - primary analysis of sensitivity comparison based on the blinded readers' assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 1; Test type: Superiority; p = 0.8694, McNemar 1-sided test,alpha level of 2.5%; Sensitivity Difference = -0.7, 95% CI 1-sided [lower limit -8.5]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 2 for presence of a myocardial perfusion defect indicating significant cad per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - primary analysis of sensitivity comparison based on the blinded readers' assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 2; Test type: Superiority; p < 0.0001, McNemar 1-sided test,alpha level of 2.5%; Sensitivity Difference = 29.1, 95% CI 1-sided [lower limit 21.7]
Statistical Analysis 3: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 3 for presence of a myocardial perfusion defect indicating significant cad per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - primary analysis of sensitivity comparison based on the blinded readers' assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 3; Test type: Superiority; p < 0.0001, McNemar 1-sided test,alpha level of 2.5%; Sensitivity Difference = 24.1, 95% CI 1-sided [lower limit 16.6]

6. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Additional Secondary Analysis of Sensitivity Comparison Based on the Blinded Readers' Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by blinded readers' assessment. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=70% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 108
Sensitivity %
  Gadobutrol-enhanced CMRI-Reader 1 | 89.8
  Gadobutrol-enhanced CMRI-Reader 2 | 79.6
  Gadobutrol-enhanced CMRI-Reader 3 | 78.7
  Unenhanced CMRI-Reader 1 | 82.4
  Unenhanced CMRI-Reader 2 | 45.4
  Unenhanced CMRI-Reader 3 | 48.1
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 1 for presence of a myocardial perfusion defect indicating significant CAD per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - additional secondary analysis of sensitivity comparison based on the blinded readers' assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 1; Test type: Superiority; p = 0.0455, McNemar 1-sided test,alpha level of 2.5%; Sensitivity Difference] = 7.4, 95% CI 1-sided [lower limit 0.5]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 2 for presence of a myocardial perfusion defect indicating significant CAD per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - additional secondary analysis of sensitivity comparison based on the blinded readers' assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 2; Test type: Superiority; p < 0.0001, McNemar 1-sided test,alpha level of 2.5%; Sensitivity Difference] = 34.3, 95% CI 1-sided [lower limit 25.2]
Statistical Analysis 3: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 3 for presence of a myocardial perfusion defect indicating significant CAD per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - additional secondary analysis of sensitivity comparison based on the blinded readers' assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 3; Test type: Superiority; p < 0.0001, McNemar 1-sided test,alpha level of 2.5%; Sensitivity Difference = 30.6, 95% CI 1-sided [lower limit 21.7]

7. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Secondary Analysis of Sensitivity Based on Investigator's Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by investigator's assessment. Significant CAD was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or the presence of wall motion abnormalities on unenhanced CMRI images verified by SoR (significant CAD defined as QCA stenosis of >=50%). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 140
Sensitivity % | 74.3 [66.2 to 81.3]

8. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Sensitivity Comparison Based on Investigator's Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by investigator's assessment. Significant CAD was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or the presence of wall motion abnormalities on unenhanced CMRI images verified by SoR (significant CAD defined as QCA stenosis of >=70%). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 108
Sensitivity % | 89.8 [82.5 to 94.8]

9. Secondary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Secondary Analysis of Specificity Based on Investigator's Assessment
Description: Investigator's assessment evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest). A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. The investigator's assessment of participant-based specificity of gadobutrol-enhanced CMRI was analyzed with significant CAD defined as maximum stenosis severity of >=50% by QCA, which were secondary analysis. Specificity= true negative/ (true negative + false positive).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 234
Specificity % | 85.9 [80.8 to 90.1]

10. Secondary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Specificity Based on Investigator's Assessment
Description: Investigator's assessment evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest). A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. The investigator's assessment of participant-based specificity of gadobutrol-enhanced CMRI was analyzed with significant CAD defined as maximum stenosis severity of >=70% by QCA, which were secondary analysis. Specificity= true negative/ (true negative + false positive). This additional secondary analysis of specificity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 266
Specificity % | 85.0 [80.1 to 89.0]

11. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Secondary Analysis of Sensitivity Comparison Based on Investigator's Assessment
Description: Investigator's assessment evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest). A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. The investigator's assessment of participant-based sensitivity and specificity of gadobutrol-enhanced CMRI was analyzed with significant CAD defined as maximum stenosis severity of >=50% by QCA, which were secondary analysis. Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 141
Sensitivity %
  Gadobutrol-enhanced CMRI | 74.3
  Unenhanced CMRI | 46.4
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 1 for presence of a myocardial perfusion defect indicating significant CAD per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - secondary analysis of sensitivity comparison based on investigator's assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI. Maximum stenosis severity at least >=50% by QCA; Test type: Superiority; p < 0.0001, McNemar 2-sided test,alpha level of 5%; Sensitivity Difference = 27.9, 95% CI 2-sided [18.5 to 35.8]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Statistical analysis 2 for presence of a myocardial perfusion defect indicating significant CAD per participant on gadobutrol-enhanced CMRI versus unenhanced wall motion CMRI images - secondary analysis of sensitivity comparison based on investigator's assessment. Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI. Maximum stenosis severity at least >=50% by QCA; Test type: Superiority; p < 0.0001, McNemar 2-sided test,alpha level of 10%; Sensitivity Difference = 27.9, 95% CI 2-sided [19.9 to 34.4]

12. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Additional Secondary Analysis of Sensitivity Comparison Based on Investigator's Assessment
Description: Investigator's assessment evaluated 6 myocardial regions based on regional perfusion score (RPS), 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest). A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. The investigator's assessment of participant-based sensitivity and specificity of gadobutrol-enhanced CMRI was analyzed with significant CAD defined as maximum stenosis severity of >=70% by QCA, which were secondary analysis. Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 108
Sensitivity %
  Gadobutrolenhanced:True Positive(Sensitivity) | 89.8
  Unenhanced: True Positive (Sensitivity) | 57.4

13. Secondary Outcome: Localization of a Myocardial Perfusion Defect to a Coronary Territory on Gadobutrol-Enhanced CMRI - Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessments
Description: Sensitivity was calculated coronary territory based, a coronary territory (left anterior descending artery [LAD] / non-LAD / right coronary artery [RCA] / left circumflex artery [LCX]) was rated positive for significant CAD (significant CAD defined as QCA stenosis of>=50%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory(LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Sensitivity was displayed for all 3 blinded readers and the investigator.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 103
Sensitivity %
  Localization to LAD territory: Reader 1: number analyzed (Participants) | 96
  Localization to LAD territory: Reader 1 | 43.8
  Localization to LAD territory: Reader 2: number analyzed (Participants) | 96
  Localization to LAD territory: Reader 2 | 31.3
  Localization to LAD territory: Reader 3: number analyzed (Participants) | 96
  Localization to LAD territory: Reader 3 | 34.4
  Localization to LAD territory: Investigator: number analyzed (Participants) | 95
  Localization to LAD territory: Investigator | 45.3
  Localization to non-LAD territory: Reader 1 | 84.5
  Localization to non-LAD territory: Reader 2 | 68.9
  Localization to non-LAD territory: Reader 3 | 71.8
  Localization to non-LAD territory: Investigator | 76.7
  Localization to RCA territory: Reader 1: number analyzed (Participants) | 76
  Localization to RCA territory: Reader 1 | 85.5
  Localization to RCA territory: Reader 2: number analyzed (Participants) | 76
  Localization to RCA territory: Reader 2 | 69.7
  Localization to RCA territory: Reader 3: number analyzed (Participants) | 76
  Localization to RCA territory: Reader 3 | 69.7
  Localization to RCA territory: Investigator: number analyzed (Participants) | 76
  Localization to RCA territory: Investigator | 71.1
  Localization to LCX territory: Reader 1: number analyzed (Participants) | 72
  Localization to LCX territory: Reader 1 | 69.4
  Localization to LCX territory: Reader 2: number analyzed (Participants) | 72
  Localization to LCX territory: Reader 2 | 48.6
  Localization to LCX territory: Reader 3: number analyzed (Participants) | 72
  Localization to LCX territory: Reader 3 | 47.2
  Localization to LCX territory: Investigator: number analyzed (Participants) | 72
  Localization to LCX territory: Investigator | 55.6

14. Secondary Outcome: Localization of a Myocardial Perfusion Defect to a Coronary Territory on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessments
Description: Sensitivity was calculated coronary territory based, a coronary territory (LAD / non-LAD / RCA / LCX) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=70%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Sensitivity was displayed for all 3 blinded readers and the investigator. This additional secondary analysis of sensitivity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 87
Sensitivity %
  Localization to LAD territory: Reader 1: number analyzed (Participants) | 51
  Localization to LAD territory: Reader 1 | 70.6
  Localization to LAD territory: Reader 2: number analyzed (Participants) | 51
  Localization to LAD territory: Reader 2 | 52.9
  Localization to LAD territory: Reader 3: number analyzed (Participants) | 51
  Localization to LAD territory: Reader 3 | 56.9
  Localization to LAD territory: Investigator: number analyzed (Participants) | 51
  Localization to LAD territory: Investigator | 68.6
  Localization to non-LAD territory: Reader 1 | 90.8
  Localization to non-LAD territory: Reader 2 | 78.2
  Localization to non-LAD territory: Reader 3 | 80.5
  Localization to non-LAD territory: Investigator | 88.5
  Localization to RCA territory: Reader 1: number analyzed (Participants) | 62
  Localization to RCA territory: Reader 1 | 90.3
  Localization to RCA territory: Reader 2: number analyzed (Participants) | 62
  Localization to RCA territory: Reader 2 | 80.6
  Localization to RCA territory: Reader 3: number analyzed (Participants) | 62
  Localization to RCA territory: Reader 3 | 82.3
  Localization to RCA territory: Investigator: number analyzed (Participants) | 62
  Localization to RCA territory: Investigator | 83.9
  Localization to LCX territory: Reader 1: number analyzed (Participants) | 48
  Localization to LCX territory: Reader 1 | 77.1
  Localization to LCX territory: Reader 2: number analyzed (Participants) | 48
  Localization to LCX territory: Reader 2 | 50.0
  Localization to LCX territory: Reader 3: number analyzed (Participants) | 48
  Localization to LCX territory: Reader 3 | 50.0
  Localization to LCX territory: Investigator: number analyzed (Participants) | 48
  Localization to LCX territory: Investigator | 70.8

15. Secondary Outcome: Localization of a Myocardial Perfusion Defect to a Coronary Territory on Gadobutrol-enhanced CMRI - Secondary Analysis of Specificity Based on Blinded Readers' and Investigator's Assessments
Description: Specificity was calculated coronary territory based, a coronary territory (LAD / non-LAD / RCA / LCX) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Specificity was displayed for all 3 blinded readers and the investigator.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 138
Specificity %
  Localization to LAD territory: Reader 1 | 92.8
  Localization to LAD territory: Reader 2 | 97.1
  Localization to LAD territory: Reader 3 | 93.5
  Localization to LAD territory: Investigator: number analyzed (Participants) | 137
  Localization to LAD territory: Investigator | 91.2
  Localization to non-LAD territory: Reader 1: number analyzed (Participants) | 86
  Localization to non-LAD territory: Reader 1 | 91.9
  Localization to non-LAD territory: Reader 2: number analyzed (Participants) | 86
  Localization to non-LAD territory: Reader 2 | 97.7
  Localization to non-LAD territory: Reader 3: number analyzed (Participants) | 86
  Localization to non-LAD territory: Reader 3 | 96.5
  Localization to non-LAD territory: Investigator: number analyzed (Participants) | 85
  Localization to non-LAD territory: Investigator | 95.3
  Localization to RCA territory: Reader 1: number analyzed (Participants) | 124
  Localization to RCA territory: Reader 1 | 82.3
  Localization to RCA territory: Reader 2: number analyzed (Participants) | 124
  Localization to RCA territory: Reader 2 | 91.1
  Localization to RCA territory: Reader 3: number analyzed (Participants) | 124
  Localization to RCA territory: Reader 3 | 87.9
  Localization to RCA territory: Investigator: number analyzed (Participants) | 122
  Localization to RCA territory: Investigator | 87.7
  Localization to LCX territory: Reader 1: number analyzed (Participants) | 108
  Localization to LCX territory: Reader 1 | 88.9
  Localization to LCX territory: Reader 2: number analyzed (Participants) | 108
  Localization to LCX territory: Reader 2 | 94.4
  Localization to LCX territory: Reader 3: number analyzed (Participants) | 108
  Localization to LCX territory: Reader 3 | 95.4
  Localization to LCX territory: Investigator: number analyzed (Participants) | 107
  Localization to LCX territory: Investigator | 93.5

16. Secondary Outcome: Localization of a Myocardial Perfusion Defect to a Coronary Territory on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Specificity Based on Blinded Readers' and Investigator's Assessments
Description: Specificity was calculated coronary territory based, a coronary territory (LAD / non-LAD / RCA / LCX) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=70%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Specificity was displayed for all 3 blinded readers and the investigator. This additional secondary analysis of specificity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 190
Specificity %
  Localization to LAD territory: Reader 1 | 90.0
  Localization to LAD territory: Reader 2 | 95.3
  Localization to LAD territory: Reader 3 | 91.1
  Localization to LAD territory: Investigator: number analyzed (Participants) | 188
  Localization to LAD territory: Investigator | 86.7
  Localization to non-LAD territory: Reader 1: number analyzed (Participants) | 98
  Localization to non-LAD territory: Reader 1 | 85.7
  Localization to non-LAD territory: Reader 2: number analyzed (Participants) | 98
  Localization to non-LAD territory: Reader 2 | 92.9
  Localization to non-LAD territory: Reader 3: number analyzed (Participants) | 98
  Localization to non-LAD territory: Reader 3 | 91.8
  Localization to non-LAD territory: Investigator: number analyzed (Participants) | 97
  Localization to non-LAD territory: Investigator | 91.8
  Localization to RCA territory: Reader 1: number analyzed (Participants) | 147
  Localization to RCA territory: Reader 1 | 74.8
  Localization to RCA territory: Reader 2: number analyzed (Participants) | 147
  Localization to RCA territory: Reader 2 | 87.1
  Localization to RCA territory: Reader 3: number analyzed (Participants) | 147
  Localization to RCA territory: Reader 3 | 85.0
  Localization to RCA territory: Investigator: number analyzed (Participants) | 145
  Localization to RCA territory: Investigator | 85.5
  Localization to LCX territory: Reader 1: number analyzed (Participants) | 141
  Localization to LCX territory: Reader 1 | 78.7
  Localization to LCX territory: Reader 2: number analyzed (Participants) | 141
  Localization to LCX territory: Reader 2 | 85.8
  Localization to LCX territory: Reader 3: number analyzed (Participants) | 141
  Localization to LCX territory: Reader 3 | 87.2
  Localization to LCX territory: Investigator: number analyzed (Participants) | 140
  Localization to LCX territory: Investigator | 87.9

17. Secondary Outcome: Detection of Myocardial Perfusion Defect(s) on Gadobutrol-enhanced CMRI in Participants With Significant LMS Stenosis - Based on Blinded Readers' and Investigator's Assessments
Description: Sensitivity was calculated for detection of myocardial perfusion defects on gadobutrol-enhanced CMRI in participants with significant left main stem (LMS) stenosis and the myocardial perfusion defect pattern was described. If >=1 myocardial region showed a myocardial perfusion defect with a RPS of >=1, participants will be rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: FAS included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for SoR diagnosis were available. N=FAS participants with significant CAD (defined as maximum stenosis severity of >=50% by QCA) as verified by SoR in the LMS.
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 9
Participants
  Isolated, Reader 1 | 1
  Single-vessel, Reader 1 | 2
  2-vessel, Reader 1 | 1
  3-vessel, Reader 1 | 3
  Isolated, Reader 2 | 0
  Single-vessel, Reader 2 | 2
  2-vessel, Reader 2 | 1
  3-vessel, Reader 2 | 3
  Isolated, Reader 3 | 0
  Single-vessel, Reader 3 | 2
  2-vessel, Reader 3 | 1
  3-vessel, Reader 3 | 3
  Isolated, Investigator | 0
  Single-vessel, Investigator | 2
  2-vessel, Investigator | 2
  3-vessel, Investigator | 3

18. Secondary Outcome: Presence/Absence of a MPD Indicating/Excluding Significant CAD in Participants With Multi Versus Single Vessel Disease Evaluated on Gadobutrol-enhanced CMRI-Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessments
Description: Sensitivity was calculated for detection of myocardial perfusion defects (MPD) on gadobutrol-enhanced CMRI in participants with single and multi-vessel diseases. If >=1 myocardial region showed a myocardial perfusion defect with a RPS of >=1, participants will be rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 75
Sensitivity %
  Single-vessel disease - Reader 1: number analyzed (Participants) | 57
  Single-vessel disease - Reader 1 | 56.1 [42.4 to 69.3]
  Single-vessel disease - Reader 2: number analyzed (Participants) | 57
  Single-vessel disease - Reader 2 | 50.9 [37.3 to 64.4]
  Single-vessel disease - Reader 3: number analyzed (Participants) | 57
  Single-vessel disease - Reader 3 | 49.1 [35.6 to 62.7]
  Single-vessel disease - Investigator: number analyzed (Participants) | 56
  Single-vessel disease - Investigator | 57.1 [43.2 to 70.3]
  Multi-vessel disease - Reader 1 | 92.0 [83.4 to 97.0]
  Multi-vessel disease - Reader 2 | 76.0 [64.7 to 85.1]
  Multi-vessel disease - Reader 3 | 76.0 [64.7 to 85.1]
  Multi-vessel disease - Investigator | 86.7 [76.8 to 93.4]

19. Secondary Outcome: Presence/Absence of a MPD Indicating/Excluding Significant CAD in Participants With Multi Vs Single Vessel Disease Evaluated on Gadobutrol-enhanced CMRI-Additional Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessments
Description: Sensitivity was calculated for detection of MPD on gadobutrol-enhanced CMRI in participants with single and multi-vessel diseases. If >=1 myocardial region showed a myocardial perfusion defect with a RPS of >=1, participants will be rated positive for significant CAD (significant CAD defined as QCA stenosis of >=70%). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was prospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 68
Sensitivity %
  Single-vessel disease - Reader 1 | 85.3
  Single-vessel disease - Reader 2 | 76.5
  Single-vessel disease - Reader 3 | 76.5
  Single-vessel disease - Investigator | 86.8
  Multi-vessel disease - Reader 1: number analyzed (Participants) | 40
  Multi-vessel disease - Reader 1 | 97.5
  Multi-vessel disease - Reader 2: number analyzed (Participants) | 40
  Multi-vessel disease - Reader 2 | 85.0
  Multi-vessel disease - Reader 3: number analyzed (Participants) | 40
  Multi-vessel disease - Reader 3 | 82.5
  Multi-vessel disease - Investigator: number analyzed (Participants) | 40
  Multi-vessel disease - Investigator | 95.0

20. Secondary Outcome: Percentage of Participants by Their Lowest Confidence in Diagnosis Obtained on Gadobutrol-enhanced CMRI and Unenhanced Wall Motion CMRI - Based on Blinded Readers' and Investigator's Assessments
Description: Score for confidence in diagnosis (not confident, somewhat confident, and confident) was described descriptively for each of the 6 myocardial regions. The frequency over the worst confidence in diagnosis obtained within a participant was displayed. All these analyses were done separately for gadobutrol-enhanced CMRI and unenhanced wall motion CMRI.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 376
Percentage of Participants
  Unenhanced/Reader 1: Confident | 74.7
  Unenhanced/Reader 1: Somewhat confident | 15.7
  Unenhanced/Reader 1: Not confident | 9.6
  Unenhanced/Reader 1: Missing | 0
  Unenhanced/Reader 2: Confident | 86.4
  Unenhanced/Reader 2: Somewhat confident | 12.8
  Unenhanced/Reader 2: Not confident | 0.8
  Unenhanced/Reader 2: Missing | 0
  Unenhanced/Reader 3: Confident | 63.0
  Unenhanced/Reader 3: Somewhat confident | 36.4
  Unenhanced/Reader 3: Not confident | 0.5
  Unenhanced/Reader 3: Missing | 0
  Unenhanced/Investi.: Confident | 91.2
  Unenhanced/Investi.: Somewhat confident | 8.2
  Unenhanced/Investi.: Not confident | 0.3
  Unenhanced/Investi.: Missing | 0.3
  Gadobutrol-enhanced/Reader 1: Confident | 88.3
  Gadobutrol-enhanced/Reader 1: Somewhat confident | 8.2
  Gadobutrol-enhanced/Reader 1: Not confident | 3.5
  Gadobutrol-enhanced/Reader 1: Missing | 0
  Gadobutrol-enhanced/Reader 2: Confident | 75.5
  Gadobutrol-enhanced/Reader 2: Somewhat confident | 23.4
  Gadobutrol-enhanced/Reader 2: Not confident | 1.1
  Gadobutrol-enhanced/Reader 2: Missing | 0
  Gadobutrol-enhanced/Reader 3: Confident | 74.7
  Gadobutrol-enhanced/Reader 3: Somewhat confident | 23.7
  Gadobutrol-enhanced/Reader 3: Not confident | 1.6
  Gadobutrol-enhanced/Reader 3: Missing | 0
  Gadobutrol-enhanced/Investi.: Confident | 79.0
  Gadobutrol-enhanced/Investi.: Somewhat confident | 19.1
  Gadobutrol-enhanced/Investi.: Not confident | 1.3
  Gadobutrol-enhanced/Investi.: Missing | 0.5

ADVERSE EVENTS:
Time Frame: From the time of gadobutrol injection until 24 ± 6 hours follow-up
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
All-Cause Mortality (participants affected / at risk) | 0/426
Serious Adverse Events (participants affected / at risk) | 1/426
Other Adverse Events (participants affected / at risk) | 47/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.1 mmol/kg Body Weight (N=426)
Chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.1 mmol/kg Body Weight (N=426)
Angina pectoris (Cardiac disorders) | 5 (6)
Bradycardia (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 10 (11)
Chest pain (General disorders) | 2 (2)
Feeling hot (General disorders) | 5 (5)
Pain (General disorders) | 1 (1)
Blood pressure decreased (Investigations) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Head discomfort (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (8)
Paraesthesia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Panic reaction (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2)
Microangiopathy (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is interested in the publication of the results of every study it performs. All relevant aspects regarding the publication will be part of the contract between the sponsor and the investigator/institution. The sponsor has made the information regarding the study protocol publicly available on the internet at www.clinicaltrials.gov.